CLINICAL TRIAL: NCT07263932
Title: Postoperative Analgesic Effectiveness of Pericapsular Nerve Block (PENG) and Posterior Hip Pericapsular Block (PHPB) in Hip Arthroplasty
Brief Title: PENG vs PHPB for Hip Arthroplasty Analgesia
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-25-12993
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: PENG Block; Hip Arthroplasty, Total; QoR-15; Numeric Rating Scale

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PENG Group: The group that will receive the preoperative Pericapsular Nerve Group (PENG) block
  Interventions: Procedure: PENG Block
- PENG + PHPB Group: The group that will receive the preoperative Pericapsular Nerve Group (PENG) block and Posterior Hip Pericapsular Block (PHPB)
  Interventions: Procedure: PENG Block and Posterior Hip Pericapsular Block

INTERVENTIONS:
Procedure: PENG Block and Posterior Hip Pericapsular Block — Patients in this group will also undergo elective total hip arthroplasty (THA) under spinal anesthesia.A preoperative Pericapsular Nerve Group (PENG) block will be performed under ultrasound guidance using 20 mL of 0.25% bupivacaine. The injection will be administered between the psoas tendon and the iliac bone to block the articular branches of the femoral, obturator, and accessory obturator nerves, providing analgesia to the anterior hip capsule. In addition to the PENG block, a Posterior Hip Pericapsular Block (PHPB) will be performed under ultrasound guidance using 20 mL of 0.25% bupivacaine. The local anesthetic will be injected between the piriformis muscle and the ischiofemoral ligament to target the posterior articular branches of the quadratus femoris, superior gluteal, and inferior gluteal nerves. The combined PENG + PHPB approach aims to provide comprehensive analgesia of both the anterior and posterior hip capsule while preserving motor function.
  Groups: PENG + PHPB Group
Procedure: PENG Block — Patients in this group will also undergo elective total hip arthroplasty (THA) under spinal anesthesia.A preoperative Pericapsular Nerve Group (PENG) block will be performed under ultrasound guidance using 20 mL of 0.25% bupivacaine. The injection will be administered between the psoas tendon and the iliac bone to block the articular branches of the femoral, obturator, and accessory obturator nerves, providing analgesia to the anterior hip capsule.
  Groups: PENG Group

SUMMARY:
Total hip arthroplasty (THA) is a commonly performed surgical procedure, and its incidence continues to rise with the aging population. Effective postoperative analgesia facilitates early mobilization and accelerates recovery. The pericapsular nerve group (PENG) block provides analgesia to the anterior hip capsule by targeting the articular branches of the femoral, obturator, and accessory obturator nerves. However, due to the contribution of sacral plexus-derived nerves (quadratus femoris, superior gluteal, and inferior gluteal nerves) to posterior hip pain, anterior blocks alone may be insufficient.

This prospective study aims to compare the efficacy of preoperatively administered PENG block alone versus the combination of PENG and posterior hip pericapsular block (PHPB) in postoperative pain control after total hip arthroplasty. The primary outcome is postoperative pain intensity assessed by the Numerical Rating Scale (NRS). Secondary outcomes include the Quality of Recovery score (QoR-15), opioid consumption, manual muscle testing (MMT) results, time to mobilization, and block-related complications.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a widely performed surgical procedure, and its incidence continues to increase with the aging population. It is an effective intervention to improve the quality of life in patients with advanced osteoarthritis or rheumatoid arthritis. Postoperative pain is one of the most common complications following THA. Effective postoperative analgesia facilitates early mobilization and accelerates recovery. Early mobilization within the first 24 hours after surgery has been shown to significantly reduce the length of hospital stay.

Regional anesthesia techniques for postoperative analgesia in hip surgery play a crucial role in pain management and recovery. International pain management guidelines recommend multimodal analgesic protocols for elective total hip arthroplasty, emphasizing the role of peripheral nerve blocks as part of these strategies.

Current anatomical studies have demonstrated that the innervation of the hip joint capsule is derived from multiple nerves originating from the lumbosacral plexus. The density and distribution of this neural supply may vary among individuals depending on pelvic morphology, ethnicity, and sex. The anterior portion of the hip joint capsule is primarily innervated by articular branches of the femoral and obturator nerves, while the posterior aspect receives innervation from branches of the sciatic nerve, the superior gluteal nerve, and the nerve to quadratus femoris (NQF). The NQF, which provides significant sensory input to the posterior hip region, has become a key anatomical target for posterior hip-focused regional anesthesia techniques.

The pericapsular nerve group (PENG) block, first described by Girón-Arango et al., provides analgesia to the anterior hip capsule by blocking the articular branches of the femoral, obturator, and accessory obturator nerves. PENG block has been suggested to facilitate early mobilization and recovery compared to other anterior approaches. However, even with appropriate anterior blocks, posterior gluteal pain may persist in patients with hip pathology. This highlights the potential importance of targeting sacral plexus-derived nerves for comprehensive analgesia.

Recent research has shown that branches from the quadratus femoris nerve (NQF), superior gluteal nerve (SGN), and inferior gluteal nerve (IGN) contribute to the posterior capsule innervation of the hip joint. Regional anesthesia techniques targeting these posterior articular branches may enhance postoperative analgesia, promote early mobilization, and improve functional recovery. Consequently, the integration of sacral plexus-focused posterior blocks alongside anterior approaches is increasingly being emphasized in multimodal analgesia protocols for THA.

The combination of the posterior hip pericapsular block (PHPB) with the PENG block has been reported to provide balanced and effective analgesia across the entire hip capsule while preserving motor function.

The aim of this prospective study is to compare the efficacy of preoperatively administered PENG block alone versus the combination of PENG and posterior hip pericapsular block (PHPB) for postoperative pain control in patients undergoing total hip arthroplasty. The primary endpoint is postoperative pain intensity assessed using the Numerical Rating Scale (NRS). Secondary endpoints include the Quality of Recovery (QoR-15) score, opioid consumption, manual muscle testing (MMT) results, time to mobilization, and block-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective total hip arthroplasty (THA) under spinal anesthesia
* ASA physical status I-II
* Age ≥18 years
* Body Mass Index (BMI) between 18-35 kg/m²
* Patients who provide written informed consent

Exclusion Criteria:

* Age <18 years
* ASA physical status ≥III
* Known allergy or contraindication to study medications (local anesthetics, opioids, etc.)
* Severe cardiac, renal, hepatic, or pulmonary failure
* Revision total hip arthroplasty
* Coagulopathy or anticoagulant use
* Local infection or neuropathic findings at the injection site
* Chronic inflammatory diseases or chronic corticosteroid use
* Diagnosed neuropsychiatric disorders
* Pregnancy or lactation
* Inability or unwillingness to read, understand, or sign the informed consent form
* Obesity (BMI >35 kg/m²)
* Failed spinal anesthesia or conversion to general anesthesia
* Active malignancy or patients receiving radiotherapy/chemotherapy
* Active systemic infection or ongoing antibiotic therapy (except prophylaxis)
* Contraindication to regional anesthesia techniques
* Chronic opioid or analgesic use for pain disorders
* History of intracranial mass, increased intracranial pressure, epilepsy, cerebrovascular accident, neuromuscular disease, or motor/sensory deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older, classified as ASA physical status I-II, scheduled for elective total hip arthroplasty under spinal anesthesia at Ankara Bilkent City Hospital. A total of 132 patients who meet the inclusion criteria and provide written informed consent will be enrolled in this single-center, prospective, randomized controlled trial.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Up to 48 hours postoperatively
  Postoperative pain will be assessed using the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain) at rest and during movement at 0, 2, 6, 8, 12, 24, 36, and 48 hours after surgery. The NRS scores will be compared between the two study groups (PENG vs. PENG + PHPB) to evaluate the effectiveness of the blocks in postoperative analgesia following total hip arthroplasty.

SECONDARY OUTCOMES:
QUALİTY OF RECOVERY-15 | Preoperative, 24, and 48 hours postoperatively
  The quality of postoperative recovery will be assessed using the validated 15-item Quality of Recovery questionnaire (QoR-15). The total score ranges from 0 (very poor recovery) to 150 (excellent recovery). The score will be measured preoperatively and at 24 and 48 hours postoperatively to compare recovery quality between the two groups.
MANUEL MUSCLE TEST | 6, 12, and 24 hours postoperatively
  Quadriceps muscle strength will be evaluated using the Manual Muscle Test (MMT) scale at 6, 12, and 24 hours after surgery. The MMT scale ranges from 0 (no contraction) to 5 (normal strength). A score <3 indicates quadriceps weakness.
Rescue analgesic | 0-48 hours postoperatively
  The time from the end of surgery to the patient's first request for rescue analgesia will be recorded. Rescue analgesia consists of intravenous tramadol 100 mg administered if the Numeric Rating Scale (NRS) score is ≥ 4. This measure will compare the analgesic duration provided by the two blocks (PENG vs. PENG + PHPB).
Postoperative Nausea and Vomiting (PONV) | 0-48 hours postoperatively
  The presence of postoperative nausea and/or vomiting will be recorded during the first 48 hours following surgery.
Length of Hospital Stay | Up to discharge (approximately 3-5 days postoperatively)
  The duration of hospitalization will be measured from the day of surgery to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulkadir But, Professor, Study Director — Ankara Bilkent City Hospital Departmant of Anesthesiology and Reanimation,Ankara,Çankaya
Locations (1):
- Ankara Bilkent City Hospital Departmant of Anesthesiology and Reanimation, Ankara,Çankaya, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Atalay YO, Ciftci B, Tekin B, Ansen G, Sakul BU, Cacan MA, Azboy I, Yilmaz B, Alici HA. A Case Series of Deep Subgluteal Block: A New Block Targeting the Missed Portion of the Hip for Analgesia After Total Hip Replacement. A A Pract. 2024 Sep 9;18(9):e01848. doi: 10.1213/XAA.0000000000001848. eCollection 2024 Sep 1. PMID 39250338
- [Result] Duan L, Li J, Chen Z, Wen T, He J, Zhang A. Posterior Hip Pericapsular Block (PHPB) with pericapsular nerve group (PENG) block for hip fracture: a case series. BMC Anesthesiol. 2024 Oct 1;24(1):352. doi: 10.1186/s12871-024-02731-2. PMID 39354374
- [Result] Vermeylen K, Van Aken D, Versyck B, Casaer S, Bleys R, Bracke P, Groen G. Deep posterior gluteal compartment block for regional anaesthesia of the posterior hip: a proof-of-concept pilot study. BJA Open. 2023 Feb 15;5:100127. doi: 10.1016/j.bjao.2023.100127. eCollection 2023 Mar. PMID 37587997